CLINICAL TRIAL: NCT04187404
Title: A Phase 1/2 Trial of a Novel Therapeutic Vaccine (EO2401) in Combination With Immune Check Point Blockade, for Treatment of Patients With Locally Advanced or Metastatic Adrenocortical Carcinoma, or Malignant Pheochromocytoma/Paraganglioma
Brief Title: A Novel Therapeutic Vaccine (EO2401) in Metastatic Adrenocortical Carcinoma, or Malignant Pheochromocytoma/Paraganglioma
Acronym: Spencer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Enterome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EOADR1-19
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Adrenocortical Carcinoma; Pheochromocytoma; Paraganglioma
Keywords: adrenocortical carcinoma; pheochromocytoma; paraganglioma
MeSH Terms: conditions — Adrenocortical Carcinoma; Pheochromocytoma; Paraganglioma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5-cohort study design (Experimental): Cohort 1:3-by-3 design of EO2401 in combination with nivolumab at standard dose. Three to 12 evaluable patients with adrenal carcinoma or progressive malignant pheochromocytoma/paraganglioma will be included depending on the safety profile of the administered treatments.
  Cohorts 2A (previously treated patients) and 2B (previously untreated patients): evaluation of EO2401in combination with nivolumab in 33 patients with adrenal carcinoma.
  Cohorts 3A (previously treated patients) and 3B (previously untreated patients) : evaluation of EO2401 combination with nivolumab in 20 patients (globally for both Cohorts 3A and 3B) with progressive malignant pheochromocytoma/ paraganglioma.
  Interventions: Biological: EO2401; Biological: Nivolumab
- randomized extension of Cohort 2A (3 arms): C2A-I (Experimental): Randomized extension of Cohort 2A (65 patients using a 4:1:1 ratio): 43 patients belonging to this extension of Cohort 2A will be treated by EO2401 and nivolumab in combination.
  Interventions: Biological: EO2401; Biological: Nivolumab
- randomized extension of Cohort 2A (3 arms): C2A-II (Experimental): 11 patients belonging to this extension of Cohort 2A will be treated by EO2401 alone.
  Interventions: Biological: EO2401
- randomized extension of Cohort 2A (3 arms): C2A-III (Active Comparator): 11 patients belonging to this extension of Cohort 2A who will be treated by nivolumab alone.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: EO2401 — Multiple dose of EO2401
  Arms: 5-cohort study design; randomized extension of Cohort 2A (3 arms): C2A-I; randomized extension of Cohort 2A (3 arms): C2A-II
Biological: Nivolumab — Multiple dose of nivolumab
  Arms: 5-cohort study design; randomized extension of Cohort 2A (3 arms): C2A-I; randomized extension of Cohort 2A (3 arms): C2A-III

SUMMARY:
This is a multicenter, Phase 1/2, First-In-Human study to assess the safety, tolerability, immunogenicity, and preliminary efficacy of EO2401 in Metastatic Adrenocortical Carcinoma, or Malignant Pheochromocytoma/Paraganglioma.

DETAILED DESCRIPTION:
EO2401 is an innovative cancer peptide therapeutic vaccine based on the homologies between Tumor Associated Antigens and microbiome-derived peptides that will be administered in combination with nivolumab to generate preliminary safety and efficacy data in patients with Metastatic Adrenocortical Carcinoma, or Malignant Pheochromocytoma/Paraganglioma.

ELIGIBILITY:
Main Inclusion Criteria:

1. For inclusion in Cohort 1 patients should have adrenocortical carcinoma(ACC), or malignant pheochromocytoma/paraganglioma (MPP), as defined below for Cohorts 2A and 3A.
2. For inclusion in Cohorts 2A and 2B patients should have histologically confirmed (at primary diagnosis) unresectable locally advanced or metastatic adrenocortical carcinoma.
3. For inclusion in Cohorts 3A and 3B patients should have histologically confirmed (at primary diagnosis) unresectable malignant (defined as metastatic disease, i.e. presence of chromaffin tissue in non-chromaffin organs) pheochromocytoma/paraganglioma, and RECIST defined progression should have been documented during a maximum of an 18-months period.
4. Patients with an age ≥ 18 years old.
5. Patients who are human leukocyte antigen (HLA)-A2 positive.
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
7. Patients with a life expectancy > 4 months as judged by their treating physician.
8. Patients with at least one measurable lesion according to RECIST 1.1.
9. Males or non-pregnant, non-lactating, females.
10. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.
11. Patients having received the information sheet and who have provided written informed consent prior to any study-related procedures.

Main Exclusion Criteria:

1. Patients treated with dexamethasone > 2 mg/day or equivalent (i.e. 13 mg/day of prednisone, or 53 mg/day of hydrocortisone) within 14 days before the first EO2401 administration, unless required to treat an adverse event.
2. Patients with prior treatment with immune check-point inhibitors
3. Patients with prior exposure to EO2401.
4. Patients treated with immunotherapy (meaning immunostimulatory or immunosuppressive therapy; beside excluded, or allowed, compounds per other inclusion/exclusion criteria specifications), radionuclide therapy, radiotherapy, cytoreductive therapy, or received treatment with any other investigational agent within 28 days before the first EO2401 administration.
5. Patients with an initial diagnosis of ACC less than 9 months from start of screening part 2.
6. Patients with ACC and any individual lesion according to RECIST 1.1 having a maximum diameter of more than 125 mm; irrespective if the lesion is proposed as a target lesion, or not, according to RECIST 1.1.
7. Patients with ACC with more than three organs involved by disease, combined with unresectable primary tumor.
8. Patients with ACC and uncontrolled hormonal secretion (according to the judgement of the treating physician).
9. Patients with MPP and uncontrolled blood pressure (according to the judgement of the treating physician).
10. Patients with abnormal laboratory values.
11. Patients with persistent Grade 3 or 4 toxicities.
12. Uncontrolled central nervous system (CNS) metastasis.
13. Other malignancy or prior malignancy with a disease-free interval of less than 3 years
14. Patients with clinically significant disease.
15. Patients with suspected autoimmune or active autoimmune disorder or known history of an autoimmune neurologic condition (e.g. Guillain-Barré syndrome).
16. Patients with history of solid organ transplantation or hematopoietic stem cell transplantation.
17. Patients with history or known presence of tuberculosis.
18. Pregnant and breastfeeding patients.
19. Patients with history or presence of human immunodeficiency virus and/or potentially active hepatitis B virus/hepatitis C virus infection.
20. Patients who have received live or attenuated vaccine therapy used for prevention of infectious diseases including seasonal (influenza) vaccinations within 4 weeks of the first dose of study drug.
21. Patients with a history of hypersensitivity to any excipient present in the pharmaceutical forms of the study treatments.
22. Patients treated with herbal remedies with immunostimulating properties or known to potentially interfere with major organ function.
23. Patients with known ongoing drug and alcohol abuse.
24. Patients with known or underlying medical or psychiatric condition that, in the Investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or AEs.
25. Patients deprived of their liberty, under protective custody, or guardship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Paillarse, Study Director — Enterome
Locations (12):
- MD Anderson Cancer Center, Houston, Texas, United States
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - Chu Lille, Lille
  - Centre Léon Bérard, Lyon
  - Assistance Publique - Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Lmu Klinikum, München
  - Universitätsklinikum Würzburg, Würzburg
- Azienda Ospedaliera Spedali Civili, Brescia, Italy
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Safety and efficacy data
Supporting Information: Study Protocol, SAP
Time Frame: Oct 2025
Access Criteria: Primary and key secondary outcomes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 safety lead-in assessed safety and tolerability of EO2401 in combination with nivolumab during 4 weeks. Evaluable patients in Cohort 1 will be assessed as part of the planned Cohorts 2A (non-randomized) and 3A, respectively. The schedule of EO2401 and nivolumab administrations are the same in Cohorts 2A (non randomized) and Cohort 3A as in Cohort 1.
Groups:
- Cohort 2A (Non-randomized): Cohort 2A includes patients (previously treated) with adrenocortical. Note, it also includes patients (previously treated) with adrenocortical carcinoma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab
- Randomized Extension of Cohort 2A (3 Arms): C2A-I: Patients with adrenocortical carcinoma belonging to this extension of Cohort 2A are treated by EO2401 and nivolumab in combination.
- Randomized Extension of Cohort 2A (3 Arms): C2A-II: Patients with adrenocortical carcinoma belonging to this extension of Cohort 2A will be treated by EO2401 alone.
- Randomized Extension of Cohort 2A (3 Arms): C2A-III: Patients with adrenocortical carcinoma belonging to this extension of Cohort 2A who will be treated by nivolumab alone.
- Cohort 2B (Non-randomized): Cohort 2B includes patients (previously untreated) with adrenocortical carcinoma.
  EO2401 in combination with nivolumab
- Cohort 3A (Non-randomized): Cohort 3A includes patients (previously treated) with progressive malignant pheochromocytoma/ paraganglioma. Note, it also includes patients (previously treated) with progressive malignant pheochromocytoma/ paraganglioma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab
- Cohort 3B (Non-randomized): Cohort 3B includes patients (previously untreated) with progressive malignant pheochromocytoma/ paraganglioma.
  EO2401 in combination with nivolumab
Period: Overall Study
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Started | 26 | 13 | 2 | 4 | 7 | 13 | 5
Started and Originally Enrolled in Cohort 1 (Safety lead-in). | 2 | 0 | 0 | 0 | 0 | 1 | 0
Completed | 26 | 13 | 2 | 4 | 7 | 13 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2A (Non-randomized): Cohort 2A includes patients (previously treated) with adrenocortical carcinoma. Note, it also includes patients (previously treated) with adrenocortical carcinoma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab.
- Randomized Extension of Cohort 2A (3 Arms): C2A-I: Patients with adrenocortical carcinoma belonging to this extension of Cohort 2A (previously treated) have been treated by EO2401 and nivolumab in combination.
- Randomized Extension of Cohort 2A (3 Arms): C2A-II: Patients with adrenocortical carcinoma belonging to this extension of Cohort 2A (previously treated) have been treated by EO2401 alone.
- Randomized Extension of Cohort 2A (3 Arms): C2A-III: Patients with adrenocortical carcinoma belonging to this extension of Cohort 2A (previously treated) have been treated by nivolumab alone.
- Cohort 2B (Non-randomized): Cohort 2B includes patients (previously untreated) with adrenocortical carcinoma. Note, it also includes patients (previously untreated) with adrenocortical carcinoma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab.
- Cohort 3B (Non-randomized): Cohort 3B includes patients (previously untreated) with progressive malignant pheochromocytoma/ paraganglioma. Note, it also includes patients (previously treated) with progressive malignant pheochromocytoma/ paraganglioma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab
- Total: Total of all reporting groups
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized) | Total
Number analyzed (Participants) | 26 | 13 | 2 | 4 | 7 | 13 | 5 | 70
Age, Continuous [Median (Full Range); unit: years] | 46 [31 to 61] | 54 [35 to 73] | 49.5 [38 to 61] | 52.5 [19 to 65] | 47 [43 to 72] | 55 [48 to 61] | 63 [36 to 64] | 51 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 0 | 3 | 7 | 4 | 4 | 46
  Male | 8 | 3 | 2 | 1 | 0 | 9 | 1 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 13 | 2 | 4 | 7 | 13 | 4 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 26 | 13 | 2 | 4 | 7 | 13 | 5 | 70
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Netherlands | 5 | 2 | 1 | 1 | 2 | 2 | 0 | 13
  United States | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Denmark | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Italy | 8 | 5 | 1 | 1 | 2 | 5 | 1 | 23
  France | 7 | 6 | 0 | 1 | 2 | 2 | 3 | 21
  Germany | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 4
  Spain | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Serious Adverse Events Assessment
Description: Incidences of treatment-emergent serious adverse events using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.
Time Frame: 46 months maximum (from baseline up to study end)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3B (Non-randomized): Cohort 3B includes patients (previously untreated) with progressive malignant pheochromocytoma/ paraganglioma. Note, it also includes patients (previously untreated) with progressive malignant pheochromocytoma/ paraganglioma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Number analyzed (Participants) | 26 | 13 | 2 | 4 | 7 | 13 | 5
Participants | 5 | 4 | 1 | 0 | 1 | 4 | 2

2. Primary Outcome: Treatment-Emergent Non-Serious Adverse Events
Description: Incidences of treatment-emergent non-serious adverse events using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.
Time Frame: 46 months maximum (from baseline up to study end)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Number analyzed (Participants) | 26 | 13 | 2 | 4 | 7 | 13 | 5
Participants | 26 | 13 | 2 | 4 | 7 | 13 | 5

3. Primary Outcome: All Cause Mortalities Assessment
Description: Incidence of death
Time Frame: 46 months maximum (from baseline up to study end)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 21 (Non-randomized): Cohort 2 includes patients (previously treated) with adrenocortical carcinoma. Note, it also includes patients (previously treated) with adrenocortical carcinoma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab
Arm/Group | Cohort 21 (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Number analyzed (Participants) | 26 | 13 | 2 | 4 | 7 | 13 | 5
Participants | 21 | 5 | 1 | 2 | 6 | 9 | 0

4. Secondary Outcome: Evaluation of Progression Free Survival
Description: Progression Free Survival according to iRECIST criteria at 6 months
Time Frame: 6 months after treatment start
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 2A (Non-randomized): Cohort 21 includes patients (previously treated) with adrenocortical carcinoma. Note, it also includes patients (previously treated) with adrenocortical carcinoma originally enrolled in Cohort 1 (safety lead-in).
  EO2401 in combination with nivolumab
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Number analyzed (Participants) | 26 | 13 | 2 | 4 | 7 | 13 | 5
months | 1.9 [1.8 to 2.3] | 1.9 [1.7 to 2.5] | 1.6 [1.2 to NA] — Insufficient number of participants with events | 1.7 [1.2 to NA] — Insufficient number of participants with events | 1.9 [1.2 to 2.7] | 5.2 [1.9 to 12.2] | 19.4 [3.9 to NA] — Insufficient number of participants with events

5. Secondary Outcome: Evaluation of Survival
Description: Overall survival, defined as the time interval from the date of first study treatment administration to the date of death due to any cause
Time Frame: 46 months maximum (from baseline up to study end)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Number analyzed (Participants) | 26 | 13 | 2 | 4 | 7 | 13 | 5
months | 11.9 [2.2 to 22.9] | NA [8.6 to NA] — Insufficient number of participants with events | NA [3.0 to NA] — Insufficient number of participants with events | NA [1.6 to NA] — Insufficient number of participants with events | 24.2 [1.2 to 33.5] | 11.4 [4.6 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

6. Secondary Outcome: Percentage of Patients With Immunogenicity Against EO2401
Description: Expansion of specific T cells comparing samples taken at baseline versus on treatment in an individual patient determining if the patient has a positive response to peptides that compose EO2401, or not. EO2401 immunogenicity is assessed by interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) (IVS and ex vivo).
Time Frame: 7 weeks after treatment start
Population: Patient is in C2A-III were treated with nivolumab only (not EO2401)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
Number analyzed (Participants) | 12 | 8 | 1 | 0 | 3 | 8 | 2
Participants | 12 | 8 | 0 | 0 | 3 | 5 | 2

ADVERSE EVENTS:
Time Frame: 46 months maximum (from baseline up to study end)
Description: Incidences of deaths and treatment-emergent AEs (Serious and Non-Serious) using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.
Arm/Group | Cohort 2A (Non-randomized) | Randomized Extension of Cohort 2A (3 Arms): C2A-I | Randomized Extension of Cohort 2A (3 Arms): C2A-II | Randomized Extension of Cohort 2A (3 Arms): C2A-III | Cohort 2B (Non-randomized) | Cohort 3A (Non-randomized) | Cohort 3B (Non-randomized)
All-Cause Mortality (participants affected / at risk) | 21/26 | 5/13 | 1/2 | 2/4 | 6/7 | 9/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/26 | 4/13 | 1/2 | 0/4 | 1/7 | 4/13 | 2/5
Other Adverse Events (participants affected / at risk) | 26/26 | 13/13 | 2/2 | 4/4 | 7/7 | 13/13 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2A (Non-randomized) (N=26) | Randomized Extension of Cohort 2A (3 Arms): C2A-I (N=13) | Randomized Extension of Cohort 2A (3 Arms): C2A-II (N=2) | Randomized Extension of Cohort 2A (3 Arms): C2A-III (N=4) | Cohort 2B (Non-randomized) (N=7) | Cohort 3A (Non-randomized) (N=13) | Cohort 3B (Non-randomized) (N=5)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2A (Non-randomized) (N=26) | Randomized Extension of Cohort 2A (3 Arms): C2A-I (N=13) | Randomized Extension of Cohort 2A (3 Arms): C2A-II (N=2) | Randomized Extension of Cohort 2A (3 Arms): C2A-III (N=4) | Cohort 2B (Non-randomized) (N=7) | Cohort 3A (Non-randomized) (N=13) | Cohort 3B (Non-randomized) (N=5)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (9) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (10) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Administration site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (5) | 9 (11) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (3)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (8) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immediate post-injection reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site erythema (General disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 2 (3) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site inflammation (General disorders) | 2 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site injury (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (3)
Injection site plaque (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 9 (26) | 6 (7) | 2 (3) | 0 (0) | 3 (3) | 6 (10) | 2 (3)
Injection site swelling (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 10 (17) | 3 (6) | 0 (0) | 0 (0) | 3 (3) | 4 (9) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric pH decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil morphology abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vein disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White coat hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04187404/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT04187404/SAP_001.pdf